CLINICAL TRIAL: NCT03161548
Title: A Phase II Study of Tongue Conservation Surgery for Advanced Oral Tongue Cancer: Induction Chemotherapy, Followed by Tongue Conservation Surgery and Postoperative Chemoradoitherapy
Brief Title: A Study of Tongue Conservation Surgery for Oral Tongue Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Diffiult patient recruitment
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201009018MB
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Tongue Cancer; Chemotherapy Effect; Surgery
MeSH Terms: conditions — Tongue Neoplasms | interventions — Induction Chemotherapy

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-comparative phase II clinical trial to assess efficacy and safety of tongue conservation treatment with sequential doxcetaxel, cisplatin and tegafur/uracil plus leucovorin (DCU) induction chemotherapy, tongue conservation surgery and postoperative CCRT in patients with advanced oral tongue cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (1):
- Induction chemotherapy (Experimental): Induction chemotherapy will be given every 21 days, with the DCU regimen, followed by tongue conservation surgery, and postoperative CCRT as indicated.
  Interventions: Drug: Induction chemotherapy; Procedure: Tongue conservation surgery; Radiation: postoperative CCRT

INTERVENTIONS:
Drug: Induction chemotherapy — All eligible subjects will receive ICT with DCU regimen every 21 days as follows:
  Docetaxel 36 mg/m2 intravenous infusion over 1 hr, followed by Cisplatin 30 mg/m2 intravenous infusion over 1 hr, on day 1 and day 8, Oral tegafur/uracil 300 mg/m2/day plus leucovorin 90 mg/day on days 1 - 14
Procedure: Tongue conservation surgery — Surgical excision of residual oral tongue tumor will be performed in 3-4 weeks after the start of the last cycle of ICT. Neck dissection will also be done as indicated.
Radiation: postoperative CCRT — Post-op CCRT will be started 4-6 weeks after surgery, with regimen as follows:
  Radiotherapy in 2 Gy once-daily fraction size, Monday to Friday, with dose up to 60 Gy (total of 30 fractions); Cisplatin 25 mg/m2 intravenously for 4 hours every week a cycle to total 6 cycles; Tegafur/uracil (UFUR) 200 mg po bid for whole course of radiotherapy

SUMMARY:
This is an open-label, non-comparative phase II clinical trial to assess efficacy and safety of tongue conservation treatment with sequential induction chemotherapy, tongue conservation surgery and postoperative concurrent chemoradiotherapy (CCRT) in patients with advanced oral tongue cancer.

DETAILED DESCRIPTION:
Surgical resection remains the most important component of standard treatment for oral tongue cancer, but may lead to profound functional impacts not effectively compensated by reconstruction surgery. The volume of tongue resection remains one key factor for the post-treatment deterioration of the functional outcomes and quality of life in large oral tongue cancer. Primary chemoradiotherapy without surgical resection has not been accepted for oral tongue cancer because of the concerns about possible poorer response and sequelae. Breast conservation treatment, by the sequential use of induction chemotherapy (ICT), limited surgical resection and chemoradiotherapy, has become a standard treatment for human breast cancer of various stages. However, similar tongue conservation treatment for advanced oral tongue cancer has not been studied in trials. Based on these data, it will be reasonable, in locally advanced (> 3 cm) resectable oral tongue cancers, to test whether ICT followed by tongue conservation surgery and postoperative CCRT can safely enhance the possibility of tongue conservation with improved post-treatment functions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological proof of squamous cell carcinoma of oral tongue
* b. cT2-4, N0-2,M0, by clinical or radiographic examinations
* Either mandibulotomy, mandibulectomy or flap reconstruction is required by standard surgical planning
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Between 20 and 70 years of age
* Adequate hematopoietic function as defined below:

Hemoglobin >= 10g/dl Absolute neutrophil count (ANC) >= 1,500/µL Platelets >= 100,000/µL

* Adequate organ function as defined below:

Total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine <= 1.5 x upper limit of normal Creatinine clearance > 50 ml/min

* Signed study-specific consent form prior to study entry

Exclusion Criteria:

* Patients received gross oral tongue tumor resection before evaluation
* Primary subsites other than oral tongue
* Histologic diagnosis other than squamous cell carcinoma
* Patient with synchronous primary cancers (within 6 months)
* Clinical or radiographic findings as below:

T1 tumors Gross invasion to mandible, tonsil or >1/3 base of tongue N3 disease or distant metastasis (M1)

* Prior head and neck chemotherapy or radiotherapy
* Prior esophageal cancer history
* Active cardiac disease defined as: unstable angina, uncontrolled arrhythmia, myocardial infarction within 6 months.
* Severe chronic obstructive pulmonary disease (COPD) requiring ≥ 3 hospitalizations over the past year
* Mental status not fit for clinical trial.
* Pregnant or breast feeding women, or women of child-bearing potential unless using a reliable and appropriate contraceptive method.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-07-18 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 2 weeks after completion of the last cycle of induction chemotherapy
  Response to induction chemotherapy

SECONDARY OUTCOMES:
Tongue conservation surgery feasibility rates | the date of surgery
  Feasibility of tongue conservation surgery
Pathological response of induction chemotherapy | 2 weeks after surgery
  Pathological evaluation of rediual tumor status
Longitudinal quality of life (QOL) | Date of recruitment, 2 weeks after ICT completion, 3 months after treatement copletion, 1 year after treatment completion
  Evaluation of QOL with the EORTC-C30 and HN35 QOL questionnaires
Oncologic results | 5 years after treatment completion
  Disease specific survival

IPD SHARING:
Plan to Share IPD: No